CLINICAL TRIAL: NCT05850728
Title: First in Human Clinical Trial of a Next Generation, Long-acting Injectable, Combination Antiretroviral Therapy Platform
Brief Title: First in Human Study of TLC-ART 101 (ACTU 2001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Rachel Bender Ignacio, Assistant Professor, School of Medicine, University of Washington
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007490; U01AI148055 (NIH)
Record Dates: First submitted 2023-03-23; First posted 2023-05-09 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Human Immunodeficiency Virus; Treatment; Antiretroviral Therapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Pharmacologically-guided adaptive design, in which the dose is increased or decreased if needed, based on results from prior participant arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- TLC-ART 101 Initial Dosage (Experimental): The arms will all receive the nanoparticle suspension of lopinavir, ritonavir, and tenofovir (TLC-ART 101). The arms are also called cohorts. The dose a participant receives will vary, depending upon the study results and the time of when they enroll in the study.
  The initial dosage administered to 4 participants will contain:
  lopinavir 15.6 mg, ritonavir 4.2 mg, and tenofovir 9.15 mg in 1.5mL of the formulation
  If the initial dose is appropriate, an additional 8 participants will be enrolled in Arm 1, for a total study size of 12 participants.
  Interventions: Drug: TLC-ART
- TLC-ART 101 Dosage 2A (Experimental): In the scenario in which the dosage in Arm 1 produces insufficient pharmacokinetics (PK), the dosage will be increased 2 fold in Arm 2A and administered to 4 participants.
  If Arm 2A shows ideal PK parameters, and additional 8 participants will be enrolled in this arm, for a total study size of 16 participants.
  Interventions: Drug: TLC-ART
- TLC-ART 101 Dosage 2B (Experimental): In the scenario in which the dosage in Arm 1 produces excessive drug levels, the dosage will be decreased by up to 2-5 fold (2-5x descending dose) and administered to 4 participants.
  If Arm 2B shows ideal PK parameters, and additional 8 participants will be enrolled in this arm, for a total study size of 16 participants.
  Interventions: Drug: TLC-ART
- TLC-ART 101 Dosage 3A (Experimental): In the scenario in which the dosage in Arm 2A produces insufficient drug levels, the dosage may be further increased by 2-fold from Arm 2A dosage (4x total dosage increase) and administered to an additional 4 participants.
  If Arm 3A shows ideal PK parameters, and additional 4 participants will be enrolled in this arm, for a total study size of 16 participants
  Interventions: Drug: TLC-ART
- TLC-ART 101 Dosage 3B (Experimental): In the scenario in which the dosage in Arm 2B produces excessive drug levels, the dosage may be further decreased further by up to 2-5-fold from Arm 2B dosage (4-10x dose decrease) and administered to 4 participants.
  If Arm 3B shows ideal PK parameters, and additional 4 participants will be enrolled in this arm, for a total study size of 16 participants
  Interventions: Drug: TLC-ART

INTERVENTIONS:
Drug: TLC-ART — TLC-ART 101 contains lopinavir, ritonavir, and tenofovir in a combination nanoparticle suspension

SUMMARY:
This study is a prospective, open-label, single-site, first-in-human study of a long-acting, injectable combination antiretroviral therapy platform, with a pharmacologically-guided adaptive design for dose escalation, de-escalation, and study duration. The study is designed to learn whether the formulation can be used as a platform for other drugs for treatment of HIV. The formulation is a drug combination nanoparticle (DCNP). The study will be conducted by UW Positive Research. The sample size for this study is 12-16. The study population consists of healthy adults without HIV. The study duration is 57 days per participant at the start of the study.

DETAILED DESCRIPTION:
This study is a prospective, open-label, single-site, first-in-human study of a long-acting, injectable combination antiretroviral therapy platform, with a pharmacologically-guided adaptive design for dose escalation, de-escalation, and study duration. The study has two primary aims as follows:

1. To characterize the plasma concentration-time course and pharmacokinetics (PK) of a single dose of the drug substances of TLC-ART 101 (lopinavir, ritonavir, and tenofovir) administered by subcutaneous injection within the drug combination nanoparticle.
2. To characterize the safety and tolerability of a single subcutaneous injection of TLC-ART 101.

There are 4 exploratory mechanistic objectives (with related endpoints) as follows:

1. To characterize the pharmacokinetics of the drug substances in human peripheral blood mononuclear cells (PBMCs)
2. To characterize the concentrations of intracellular TFV-diphosphate (the active moiety of TFV) in PBMCs
3. To explore whether the pharmacokinetic parameters of the 3 drug substances differ by sex following a single dose
4. To compare lymphoid tissue mononuclear cell versus PBMC concentrations of the drug substances in TLC-ART 101.

ELIGIBILITY:
Inclusion Criteria:

* Healthy with a BMI between 18.5 to 29.9 kg/m2
* Non-smoker or former smoker (defined as no smoking or no vaping or no use of tobacco cessation products for greater than 1 year)
* Persons of any gender are eligible if they otherwise meet all other entry criteria.
* Assessed by the study staff as being at low risk for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure until after completing the study.
* Willing and able to give informed consent.
* If participating in sexual activity that could lead to pregnancy, individuals of reproductive potential must agree to use specific forms of contraception throughout the study. At least two of the following must be used throughout the study:
* Condom (male or female)
* Diaphragm or cervical cap
* Copper-based intrauterine device
* Vasectomy in the male partner

Note: Select participants will have a 72-hour in-patient stay at UW Medical Center.

Note: Select participants will undergo an inguinal lymph node biopsy.

Exclusion Criteria:

Note the following criteria refer to values from the screening visit

* Positive HIV-1 fourth generation antigen/antibody test
* Positive hepatitis B surface antigen test
* Active HCV infection Note: Participants that are positive for HCV antibody must have a negative HCV RNA
* Any chronic medical condition deemed significant by the investigator (e.g., asthma, severe allergies, hypertension, heart disease, diabetes mellitus, hyperlipidemia)
* Taking any chronic oral or systemic prescription medications (including indwelling hormonal implants or hormone-releasing intrauterine devices) within 30 days before the Entry visit
* Taking any chronic oral or systemic non-prescription (over the counter, OTC) medications that cannot be safely stopped
* Any clinically significant abnormal value of CBC, creatinine, AST, ALT, alkaline phosphatase, total bilirubin
* PT/INR, PTT above the upper limit of normal
* U/A with any clinically significant abnormality
* Any clinically significant finding on ECG per physician review
* Urine toxicology screen positive for any illicit drug (other than cannabis if the participant agrees to stop use of cannabis for 14 days prior to entering the study and for the duration of the study, and is believed to be credible in this promise in the opinion of the investigator)
* BP > 140 systolic or > 90 diastolic mmHg
* Known allergy/sensitivity or any hypersensitivity to LPV, RTV, TFV or either of the lipids in TLC-ART 101 (including anaphylaxis to a COVID-19 mRNA vaccine)
* Active drug or alcohol use or dependence or psychiatric illness that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Acute or serious illness requiring systemic treatment, antibiotics, and/or hospitalization within 90 days prior to study entry
* Scars or tattoos on the central abdomen that would interfere with administration of a subcutaneous injection or assessment of the location where the study medication is planned to be administered (within 1 inch of the umbilicus)
* Diagnosis of syphilis, gonorrhea or chlamydia in the past year
* People who are pregnant, intend to become pregnant, or are breastfeeding

Additional Exclusion Criteria for Participants who will Undergo Lymph Node Biopsy

* Allergy to lidocaine or any related "-caine" drug
* Chronic scars or tattoos in both inguinal areas that might interfere with performance of a lymph node biopsy or increase the likelihood of a poor cosmetic result
* Anxiety or any other condition that has a high likelihood of interfering with the successful performance of a lymph node biopsy done under local anesthesia
* Any coagulopathy or condition that would increase the potential for bleeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Co-primary pharmacokinetic outcome: Peak TLC-101 drug substance concentrations (Cmax) in plasma | duration of follow-up in days for this study (anticipated to be 57 days per participant)
  The maximum drug substance plasma concentrations of lopinavir, ritonavir, and tenofovir obtained following a single administration
Co-primary pharmacokinetic outcome: Time to maximum TLC-101 concentration (Tmax) of drug substances in plasma | duration of follow-up in days for this study (anticipated to be 57 days per participant)
  Time taken to reach the maximum concentrations of lopinavir, ritonavir, and tenofovir over the timecourse after a single administration
Co-primary pharmacokinetic outcome: Total TLC-101 drug substance exposure (area under the curve or AUC) in plasma | duration of follow-up in days for this study (anticipated to be 57 days per participant)
  Area under the curve of plasma concentrations of lopinavir, ritonavir, and tenofovir over the study timecourse after a single administration
Co-primary pharmacokinetic outcome: Half-life (T 1/2) of TLC-101 drug substance concentrations in plasma | duration of follow-up in days for this study (anticipated to be 57 days per participant)
  The half-life of drug substance plasma concentrations of lopinavir, ritonavir, and tenofovir after a single administration
Primary safety outcome | 57 days of study follow-up, or if reported subsequent to study completion
  Treatment emergent adverse events related to TLC-ART 101 as graded by the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (Corrected Version 2.1 - July 2017)

SECONDARY OUTCOMES:
Secondary pharmacokinetic outcome: Comparison of TLC-101 drug substance concentrations in peripheral blood mononuclear cells compared with plasma levels | duration of follow-up in days for this study (anticipated to be 57 days per participant)
  To characterize the concentrations of the three drug substances in human peripheral blood mononuclear cells from the same blood samples as plasma analyses
Secondary outcome of tenofovir active drug moiety | 57 days of study follow-up
  To characterize the concentrations of intracellular tenofovir-diphosphate (the active moiety of TFV) in peripheral blood mononuclear cells
TLC-101 concentrations in lymphoid tissues | 57 days of study follow-up
  To compare lymphoid tissue mononuclear cell versus peripheral blood mononuclear cell concentrations of the drug substances in TLC-ART 101

CONTACTS AND LOCATIONS:
Overall Officials: Rachel A Bender Ignacio, MD MPH, Principal Investigator — University of Washington
Locations (1):
- UW Positve Research, Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Once study is completed, reasonable request for de-identified datasets may be considered by the study PI and sponsor
Supporting Information: Study Protocol
Time Frame: 2025-2026

REFERENCES:
- [Background] Freeling JP, Koehn J, Shu C, Sun J, Ho RJ. Anti-HIV drug-combination nanoparticles enhance plasma drug exposure duration as well as triple-drug combination levels in cells within lymph nodes and blood in primates. AIDS Res Hum Retroviruses. 2015 Jan;31(1):107-14. doi: 10.1089/aid.2014.0210. PMID 25402233
- [Background] McConnachie LA, Kinman LM, Koehn J, Kraft JC, Lane S, Lee W, Collier AC, Ho RJY. Long-Acting Profile of 4 Drugs in 1 Anti-HIV Nanosuspension in Nonhuman Primates for 5 Weeks After a Single Subcutaneous Injection. J Pharm Sci. 2018 Jul;107(7):1787-1790. doi: 10.1016/j.xphs.2018.03.005. Epub 2018 Mar 13. PMID 29548975
- [Background] Kraft JC, McConnachie LA, Koehn J, Kinman L, Collins C, Shen DD, Collier AC, Ho RJ. Long-acting combination anti-HIV drug suspension enhances and sustains higher drug levels in lymph node cells than in blood cells and plasma. AIDS. 2017 Mar 27;31(6):765-770. doi: 10.1097/QAD.0000000000001405. PMID 28099191
- [Background] Kraft JC, Treuting PM, Ho RJY. Indocyanine green nanoparticles undergo selective lymphatic uptake, distribution and retention and enable detailed mapping of lymph vessels, nodes and abnormalities. J Drug Target. 2018 Jun-Jul;26(5-6):494-504. doi: 10.1080/1061186X.2018.1433681. Epub 2018 Feb 12. PMID 29388438
- [Background] Perazzolo S, Shireman LM, McConnachie LA, Koehn J, Kinman L, Lee W, Lane S, Collier AC, Shen DD, Ho RJY. Integration of Computational and Experimental Approaches to Elucidate Mechanisms of First-Pass Lymphatic Drug Sequestration and Long-Acting Pharmacokinetics of the Injectable Triple-HIV Drug Combination TLC-ART 101. J Pharm Sci. 2020 May;109(5):1789-1801. doi: 10.1016/j.xphs.2020.01.016. Epub 2020 Jan 29. PMID 32006525
- [Background] Perazzolo S, Shireman LM, Shen DD, Ho RJY. Physiologically Based Pharmacokinetic Modeling of 3 HIV Drugs in Combination and the Role of Lymphatic System after Subcutaneous Dosing. Part 1: Model for the Free-Drug Mixture. J Pharm Sci. 2022 Feb;111(2):529-541. doi: 10.1016/j.xphs.2021.10.007. Epub 2021 Oct 19. PMID 34673093
- [Background] Perazzolo S, Shen DD, Ho RJY. Physiologically Based Pharmacokinetic Modeling of 3 HIV Drugs in Combination and the Role of Lymphatic System after Subcutaneous Dosing. Part 2: Model for the Drug-combination Nanoparticles. J Pharm Sci. 2022 Mar;111(3):825-837. doi: 10.1016/j.xphs.2021.10.009. Epub 2021 Oct 19. PMID 34673094
- See also: TLC ART Program homepage — https://depts.washington.edu/tlcart/
- See also: UW Positive Research website — https://www.uwactu.com/